CLINICAL TRIAL: NCT04960202
Title: AN INTERVENTIONAL EFFICACY AND SAFETY, PHASE 2/3, DOUBLE-BLIND, 2-ARM STUDY TO INVESTIGATE ORALLY ADMINISTERED PF-07321332/RITONAVIR COMPARED WITH PLACEBO IN NONHOSPITALIZED SYMPTOMATIC ADULT PARTICIPANTS WITH COVID-19 WHO ARE AT INCREASED RISK OF PROGRESSING TO SEVERE ILLNESS
Brief Title: EPIC-HR: Study of Oral PF-07321332/Ritonavir Compared With Placebo in Nonhospitalized High Risk Adults With COVID-19
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C4671005; 2021-002895-38 (EudraCT Number); EPIC-HR (Other: Alias Study Number)
Record Dates: First submitted 2021-07-10; First posted 2021-07-13 (Actual); Results first posted 2023-02-09 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: COVID-19
Keywords: severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2)
MeSH Terms: conditions — COVID-19 | interventions — nirmatrelvir; Ritonavir

STUDY DESIGN:
Intervention Model Description: Eligible participants with a confirmed diagnosis of SARS-CoV-2 infection will be randomized (1:1) to receive PF-07321332/ritonavir or placebo orally every 12 hours for 5 days (10 doses total).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- PF-07321332/ritonavir (Experimental): Orally administered PF-07321332+ritonavir
  Interventions: Drug: PF-07321332; Drug: Ritonavir
- Placebo (Placebo Comparator): Orally administered placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PF-07321332 — PF-07321332 (tablet)
  Arms: PF-07321332/ritonavir
Drug: Ritonavir — Ritonavir (capsule)
  Arms: PF-07321332/ritonavir
Drug: Placebo — Placebo (tablet or capsule)
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether PF-07321332/ritonavir is safe and effective for the treatment of adults who are ill with COVID-19 and do not need to be in the hospital, but are at an increased risk of developing severe illness. Throughout the study period, provision will be made to allow study visits to be conducted at a participant's home or another non-clinic location if available. The total study duration is up to 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed SARS-CoV-2 infection within 5 days prior to randomization
* Initial onset of COVID-19 signs/symptoms within 5 days prior to the day of randomization and at least 1 of the specified COVID-19 signs/symptoms present on the day of randomization
* Fertile participants must agree to use a highly effective method of contraception
* Has at least 1 characteristic or underlying medical condition associated with an increased risk of developing severe illness from COVID-19

Exclusion Criteria:

* History of or need for hospitalization for the medical treatment of COVID-19
* Prior to current disease episode, any confirmed SARS-CoV-2 infection
* Known medical history of active liver disease
* Receiving dialysis or have known moderate to severe renal impairment
* Known human immunodeficiency virus (HIV) infection with a viral load greater than 400 copies/mL or taking prohibited medications for HIV treatment
* Suspected or confirmed concurrent active systemic infection other than COVID-19
* History of hypersensitivity or other contraindication to any of the components of the study intervention
* Current or expected use of any medications or substances that are highly dependent on CYP3A4 for clearance or are strong inducers of CYP3A4
* Has received or is expected to receive convalescent COVID-19 plasma
* Has received or is expected to receive any dose of a SARS-CoV-2 vaccine before the Day 34 visit
* Participating in another interventional clinical study with an investigational compound or device, including those for COVID-19 through the long-term follow-up visit
* Known prior participation in this trial or other trial involving PF-07321332
* Oxygen saturation of <92% on room air, or on their standard home oxygen supplementation for those who regularly receive chronic supplementary oxygen for an underlying lung condition
* Females who are pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2091 (Actual)
Dates: Start 2021-07-16 (Actual); Primary Completion 2021-12-09 (Actual); Study Completion 2022-04-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (201):
- United States (73):
  - Cahaba Research Inc, Pelham, Alabama
  - The Institute for Liver Health dba Arizona Clinical Trials, Mesa, Arizona
  - The Institute for Liver Health dba Arizona Clinical Trials, Tucson, Arizona
  - Hope Clinical Research, Canoga Park, California
  - Ascada Research, Fullerton, California
  - Atella Clinical Research LLC., La Palma, California
  - Ark Clinical Research, Long Beach, California
  - American Institute of Research, Los Angeles, California
  - South Bay Clinical Research Institute, Redondo Beach, California
  - Hope Clinical Research (COVID Satellite Site), West Hills, California
  - Future Innovative Treatments, LLC, Colorado Springs, Colorado
  - Xera Med Research, Boca Raton, Florida
  - MOORE Clinical Research, Inc., Brandon, Florida
  - Innovative Research of West Florida, Inc., Clearwater, Florida
  - Herco Medical and Research Center Inc, Coral Gables, Florida
  - Advance Clinical Research Group, Cutler Bay, Florida
  - Beautiful Minds Clinical Research Center, Cutler Bay, Florida
  - Qway Research, Hialeah, Florida
  - Eastern Research Inc, Hialeah, Florida
  - Inpatient Research Clinic, Hialeah, Florida
  - Doral Medical Research LLC., Hialeah, Florida
  - Doral Medical Research,LLC, Hialeah, Florida
  - Unlimited Medical Research Group, LLC, Hialeah Gardens, Florida
  - Advanced Pulmonary Research Institute, Loxahatchee Groves, Florida
  - Angels Clinical Research Institute, Miami, Florida
  - LCC Medical Research Institute, LLC, Miami, Florida
  - Premium Medical Research Corp, Miami, Florida
  - Global Health Clinical Trials Corp, Miami, Florida
  - South Florida Research Center, Inc., Miami, Florida
  - Suncoast Research Group, LLC, Miami, Florida
  - I.V.A.M. Clinical & Investigational Center, LLC, Miami, Florida
  - C'A Research, Miami, Florida
  - ProLive Medical Research, Corp., Miami, Florida
  - Entrust Clinical Research, Miami, Florida
  - Reed Medical Research, Miami, Florida
  - Kendall South Medical Center, Miami, Florida
  - Clinical Site Partners, Inc d/b/a CSP Miami, Miami, Florida
  - Coral Research Clinic Corp, Miami, Florida
  - Savin Medical Group, LLC, Miami Lakes, Florida
  - Omega Research Orlando, LLC, Orlando, Florida
  - NAPA Research LLC, Pompano Beach, Florida
  - CDC Research Institute, Port Saint Lucie, Florida
  - USPA Advance Concept Medical Research Group LLC, South Miami, Florida
  - GCP, Global Clinical Professionals, St. Petersburg, Florida
  - Sunrise Research Institute, Sunrise, Florida
  - Santos Research Center, CORP, Tampa, Florida
  - Clinical Site Partners, Inc. dba CSP Orlando, Winter Park, Florida
  - Research by Design, LLC, Chicago, Illinois
  - New Orleans Sinus Center (COVID-19 Testing), Marrero, Louisiana
  - Tandem Clinical Research GI, LLC, Marrero, Louisiana
  - Mercury Street Medical Group, PLLC, Butte, Montana
  - Excel Clinical research, Las Vegas, Nevada
  - Meridian Clinical Research, LLC, Endwell, New York
  - Monroe Biomedical Research, Monroe, North Carolina
  - Accellacare, Wilmington, North Carolina
  - Premier Medical Group, Clarksville, Tennessee
  - PharmaTex Research, LLC, Amarillo, Texas
  - ARC Clinical Research at William Cannon, Austin, Texas
  - St Hope Foundation, Bellaire, Texas
  - Conroe Willis Medical Research, Conroe, Texas
  - South Texas Clinical Research, Corpus Christi, Texas
  - SignatureCare Emergency Center, Houston, Texas
  - Trio Clinical Trials, LLC, Houston, Texas
  - C & R Research Services USA, Houston, Texas
  - Next Level Urgent Care, Houston, Texas
  - SMS Clinical Research, LLC, Mesquite, Texas
  - SMS Clinical Research, Mesquite, Texas
  - LinQ Research, LLC, Pearland, Texas
  - Epic Medical Research, Red Oak, Texas
  - Sun Research Institute, San Antonio, Texas
  - BFHC Research, San Antonio, Texas
  - Tranquility Research, Webster, Texas
  - TPMG (Tidewater Physicians Multispecialty Group) Clinical Research, Newport News, Virginia
- Argentina (2):
  - Instituto de Investigaciones Clinicas Zarate, Zárate, Buenos Aires
  - Hospital De Clínicas Presidente Dr.Nicolas Avellaneda, San Miguel de Tucumán, Tucumán Province
- Brazil (3):
  - Chronos Pesquisa Clinica, Brasília, Federal District
  - Hospital Agamenon Magalhaes, Recife, Pernambuco
  - CECIP JAÚ - Centro de Estudos Clínicos do Interior Paulista - LTDA, Jaú, São Paulo
- Bulgaria (24):
  - Individual Practice for Primary Medical Care - IPPMC - Dr. P. Panayotov EOOD, Burgas
  - "Specialized Hospital for Active Treatment of Pneumo-Phthisiatric Diseases-Haskovo" Ltd, Haskovo
  - MHAT "Sv.Ivan. Rilski'' Kozloduy EOOD, Kozloduy
  - Diagnostic-Consultative Center I Lom EOOD, Lom
  - Multiprofile Hospital for Active Treatment- Sveti Nikolay Chudotvoretz EOOD, Lom
  - Medical centre Leo Clinic EOOD, Lovech
  - MHAT Heart and Brain EAD, Pleven
  - DCC Sveti Georgi EOOD, Plovdiv
  - MHAT "St. Panteleimon "- Plovdiv, Plovdiv
  - Multiprofile Hospital for Active Treatment Sveti Ivan Rilski - Razgrad AD, Razgrad
  - "Specialized Hospital for Active Treatment of Pneumo-Physiatric Diseases Dr. Dimitar Gramatikov -, Rousse
  - UMHAT Medica Ruse OOD, Rousse
  - Multiprofile Hospital for Active Treatment - Samokov EOOD, Samokov
  - Medical Center-1-Sevlievo EOOD, Sevlievo
  - Multiprofile Hospital For Active Treatment Shumen AD, Shumen
  - Multiprofile hospital for active treatment - Sliven to Military Medical Academy, Sliven
  - MHAT "Dr. Ivan Seliminski" AD, Sliven, Sliven
  - Diagnostic-Consultative Center XXII- Sofia ЕООD, Sofia
  - MHAT "St. Sofia" EOOD, Sofia
  - Specialized hospital for active treatment in pulmonology and phthisiology "Stara Zagora" EOOD, Stara Zagora
  - Multiprofile Hospital for Active Treatment Targovishte AD, Targovishte
  - Outpatient Clinic for Primary Outpatient Medical Care "Puls" - Dr. Mladen Buchvarov EOOD, Tsarevo
  - Medical center Leo Clinic EOOD, Varna
  - Specialized Hospital for Active Treatment of Pneumo-Phthisiatric Diseases Vratsa EOOD, Vratsa
- Fundacion Cardiomet Cequin, Armenia, Quindío Department, Colombia
- Czechia (2):
  - Zdraví-Fit, s.r.o., Protivín
  - Nemocnice Slany, Slaný
- Hungary (5):
  - Trial Pharma Kft., Békéscsaba
  - Debreceni Egyetem Klinikai Kozpont Infektologiai Klinika, Debrecen
  - Agria-Study Kft., Eger
  - Trial Pharma Kft., Gyula
  - Medifarma-98 Kft., Nyíregyháza
- India (12):
  - AIIMS Raipur, Raipur, Chhattisgarh
  - Jupiter Hospital, Vadodara, Gujarat
  - BGS Global Institute of Medical Sciences and Hospital, Bangalore, Karnataka
  - Lisie Hospital, Kochi, Kerala
  - Jehangir Clinical Development Centre Pvt. Ltd, Pune, Maharashtra
  - Lifepoint Research LLP, Pune, Maharashtra
  - Jawahar Lal Nehru Medical College, Ajmer, Rajasthan
  - Apex Hospitals Pvt Ltd, Jaipur, Rajasthan
  - Maharaja Agrasen Superspeciality Hospital, Jaipur, Rajasthan
  - Nil Ratan Sircar Medical College and Hospital, Kolkata, West Bengal
  - Aakash Healthcare Private Limited, New Delhi
  - Sardar Patel Medical College, Pavan PURI Bikaner, Rajasthan
- Japan (5):
  - International University of Health and Welfare Narita Hospital, Narita, Chiba
  - National Hokkaido Medical Center, Sapporo, Hokkaido
  - Rinku General Medical Center, Izumisano, Osaka
  - Tokyo Medical University Hachioji Medical Center, Hachiōji, Tokyo
  - National Center for Global Health and Medicine, Shinjuku, Tokyo
- Malaysia (2):
  - Hospital Umum Sarawak, Kuching, Sarawak
  - Hospital Miri, Miri, Sarawak
- Mexico (16):
  - Clinical Research Institute Saltillo S.A. de C.V., Saltillo, Coahuila
  - Asociacion Mexicana para la Investigacion Clinica A.C. (AMIC), Pachuca, Hidalgo
  - Instituto Jalisciense de Metabolismo, S.C., Guadalajara, Jalisco
  - JM Research SC, Cuernavaca, Morelos
  - Christus - Latam Hub Center of Excellence and Innovation Center S.C., Monterrey, Nuevo León
  - Eukarya Pharmasite S.C., Monterrey, Nuevo León
  - Oaxaca Site Management Organization, Oaxaca City, Oaxaca
  - InfectoLab Consultorios de Especialidad en Infectologia, Baja California, Tijuana
  - EME RED Hospitalaria, Mérida, Yucatán
  - Kohler & Milstein Research S.A. de C.V., Mérida, Yucatán
  - Centro de Investigacion Clinica Del Pacifico SA de CV, Acapulco
  - Hospital Cardiologica Aguascalientes, Aguascalientes
  - Instituto de Investigaciones Clínicas para la Salud, Durango
  - FAICIC S. de R.L. de C.V., Veracruz
  - Sociedad de Metabolismo y Corazon S.C., Veracruz
  - Arké SMO S.A de C.V, Veracruz
- Poland (2):
  - KLIMED Marek Klimkiewicz, Bialystok
  - Centrum Badań Klinicznych Piotr Napora Lekarze Spółka Partnerska, Wroclaw
- Puerto Rico (2):
  - Clinical Research Management Group Inc, Ponce
  - Advance Medical Research Center, San Juan
- Russia (4):
  - LLC Trekhgorka Medicine, Odintsovo, Moscow Oblast
  - Barnaul City Hospital Number 5, Barnaul
  - KDC "Evromedservis", OJSC, Moscow
  - Smolensk State Medical University, Smolensk
- South Africa (6):
  - MERC Welkom, Welkom, Free State
  - East Rand Research Centre T/A Worthwhile Clinical Trials, Benoni, Gauteng
  - Botho Ke Bontle Health Services, Pretoria, Gauteng
  - Synapta Clinical Research Center, Durban, KwaZulu-Natal
  - Limpopo Clinical Research Initiative, Thabazimbi, Limpopo
  - MERC Middelburg, Middelburg, Mpumalanga
- South Korea (4):
  - Kyungpook National University Chilgok Hospital, Daegu
  - Incheon Medical Center, Incheon
  - Chonnam National University Bitgoeul Hospital, Nam-gu
  - SMG-SNU Boramae Medical Center, Seoul
- Spain (2):
  - Eba Centelles, Centelles, Barcelona [barcelona]
  - Complexo Hospitalario Universitario da Coruna, A Coruña
- Thailand (6):
  - Bangkok Centre Hotel, Bang Rak, Bangkok
  - Chula Field Hospital, Chulalongkorn University Sport center (Chantanayingyong Gymnasium), Pathum Wan District,, Bangkok
  - Thai Red Cross Emerging Infectious Diseases (EDI) Clinic, Pathumwan,, Bangkok
  - The HIV Netherlands Australia Thailand Research Collaboration (HIV-NAT),, Pathumwan, Bangkok
  - Faculty of Medicine - Khon Kaen University, Muang, Changwat Khon Kaen
  - Department of Internal Medicine, Faculty of Medicine, Prince of Songkla University,, Hat Yai, Changwat Songkhla
- Turkey (Türkiye) (15):
  - Ankara University Medical Faculty, Ibni-Sina Hospital, Ankara
  - Hacettepe University Medical Faculty Hospital, Ankara
  - Akdeniz Universitesi Hastanesi, Antalya
  - Istanbul Medipol University Clinical Research Ethics Committee, Beykoz / Istanbul
  - Gaziantep University Medical Faculty, Gaziantep
  - Istanbul Yedikule Gogus Hastaliklari ve Gogus Cerrahisi Egitim Arastirma Hastanesi, Istanbul
  - Istanbul University Cerrahpasa-Cerrahpasa Medical Faculty, Istanbul
  - Acibadem Saglik Hizmetleri ve Tic.A.S, Acibadem Atakent Hastanesi, Istanbul
  - Istanbul Universitesi Klinik Arastirmalar Mukemmeliyet Uygulama ve Arastirma Merkezi, Istanbul
  - Basaksehir Cam ve Sakura Sehir Hastanesi, Istanbul
  - Kocaeli University Medical Faculty, Kocaeli
  - Sbü Dr. Suat Seren Göğüs Hastaliklari Ve Cerrahisi Eğitim Ve Araştirma Hastanesi, Konak/Izmir
  - Mersin University Health Research and Application Hospital, Mersin
  - Sakarya University Training and Research Hospital, Sakarya
  - Karadeniz Teknik Universitesi Farabi Hastanesi, Trabzon
- Ukraine (15):
  - Communal non-profit enterprise "City Clinical Hospital #16" of Dnipro City Council, Dnipro
  - Municipal Nonprofit Enterprise "Ivano-Frankivsk Regional Clinical Infectious Diseases Hospital of, Ivano-Frankivsk
  - Communal nonprofit enterprise "Central City Clinical Hospital of Ivano-Frankivsk City Council", Ivano-Frankivsk
  - Municipal Nonprofit Enterprise "City Student Hospital" of Kharkiv City Council, Kharkiv
  - Municipal Nonprofit Enterprise of Kharkiv Regional Council "Regional Clinical Infectious Diseases, Kharkiv
  - "Municipal Non-Profit Enterprise "Alexander Clinical Hospital of Kyiv" of the Kyiv City Council, Kyiv
  - Municipal non-commercial enterprise "Kyiv City Clinical Hospital #1" Of Executive Body Of the Kyiv, Kyiv
  - Kyiv Railway Clinical Hospital No.2 of Branch "Health Center of the Public Joint Stock Company, Kyiv
  - Polyclinic of Center for Medical Services and Rehabilitation of State Joint-Stock Holding Company, Kyiv
  - Municipal NonProfit Enterprise of the Lviv Regional Council Lviv Regional Information and Analitical, Lviv
  - Municipal Nonprofit Enterprise "Lviv City Clinic Hospital #4", Lviv
  - Municipal Enterprise "Poltava Regional Clinical Infectious Diseases Hospital" of Poltava Regional, Poltava
  - Municipal Enterprise "Volyn Regional Clinical Hospital" of Volyn Regional Council, Tarasove Village
  - Municipal Non-commercial Enterprise "Vinnytsia City Clinical Hospital №1", Vinnytsia
  - Communal Enterprise "Hospital #1" of Zhytomyr City Council, Zhytomyr

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Ansari W, Coetzer H, Gebo KA, Ren J, Scott A, Cappelleri JC, Cha-Silva AS, Leister-Tebbe H. Patient-Reported Outcomes of Nirmatrelvir Treatment for High-Risk, Nonhospitalized Adults With Symptomatic COVID-19. Open Forum Infect Dis. 2025 Aug 1;12(8):ofaf449. doi: 10.1093/ofid/ofaf449. eCollection 2025 Aug. PMID 40809391
- [Derived] Baniecki ML, Guan S, Rai DK, Yang Q, Lee JT, Hao L, Weinstein E, Hyde C, Cardin RD, Soares H, Hammond J. Integrated virologic analysis of resistance to nirmatrelvir/ritonavir in individuals across four phase 2/3 clinical studies for the treatment of COVID-19. EBioMedicine. 2025 Aug;118:105819. doi: 10.1016/j.ebiom.2025.105819. Epub 2025 Jun 30. PMID 40592258
- [Derived] Hammond J, Leister-Tebbe H, Gardner A, Abreu P, Bao W, Wisemandle W, Ansari W, Harrington MA, Simon-Campos A, Chew KW, Pypstra R, Rusnak JM. Alleviation of COVID-19 Symptoms and Reduction in Healthcare Utilization Among High-risk Patients Treated With Nirmatrelvir/Ritonavir (NMV/R): A Phase 3 Randomized Trial. Clin Infect Dis. 2025 Feb 24;80(2):323-330. doi: 10.1093/cid/ciae551. PMID 39523543
- [Derived] Hammond J, Leister-Tebbe H, Gardner A, Abreu P, Bao W, Wisemandle W, Baniecki M, Hendrick VM, Damle B, Simon-Campos A, Pypstra R, Rusnak JM; EPIC-HR Investigators. Oral Nirmatrelvir for High-Risk, Nonhospitalized Adults with Covid-19. N Engl J Med. 2022 Apr 14;386(15):1397-1408. doi: 10.1056/NEJMoa2118542. Epub 2022 Feb 16. PMID 35172054
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4671005

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 2256 participants signed the informed consent form (ICF). Out of these 2256 participants, 130 were screen failures who did not meet the study criteria and were not enrolled. There were 13 participants who were not screen failure but not randomized due to withdrew consent or other reasons. Of the 2113 randomized subjects, only 2091 received study treatment.
Groups:
- PF-07321332 300 mg + Ritonavir 100 mg: Participants with severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection received 300 milligrams (mg) PF-07321332 coadministered with 100 mg ritonavir orally, q12h for 5 days. Participants were followed up for safety up to Day 34 and long-term safety follow up was up to Week 24.
- Placebo: Participants with SARS-CoV-2 infection received placebo orally, q12h for 5 days. Participants were followed up for safety up to Day 34 and long-term safety follow up was up to Week 24.
Period: Overall Study
Arm/Group | PF-07321332 300 mg + Ritonavir 100 mg | Placebo
Started | 1038 | 1053
Completed | 976 | 979
Not Completed | 62 | 74
Not completed — Other | 5 | 0
Not completed — Withdrawal by Subject | 37 | 43
Not completed — Lost to Follow-up | 20 | 16
Not completed — Death | 0 | 15

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all participants randomly assigned to study intervention, whether or not administered the study intervention.
Groups:
- Total: Total of all reporting groups
Arm/Group | PF-07321332 300 mg + Ritonavir 100 mg | Placebo | Total
Number analyzed (Participants) | 1038 | 1053 | 2091
Age, Continuous [Mean (Standard Deviation); unit: Years] | 44.86 (15.37) | 45.96 (15.56) | 45.84 (15.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 522 | 515 | 1037
  Male | 516 | 538 | 1054
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 425 | 439 | 864
  Not Hispanic or Latino | 608 | 607 | 1215
  Unknown or Not Reported | 5 | 7 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 95 | 94 | 189
  Asian | 153 | 156 | 309
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 52 | 35 | 87
  White | 728 | 756 | 1484
  More than one race | 1 | 2 | 3
  Unknown or Not Reported | 9 | 10 | 19

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Covid-19 Related Hospitalization or Death From Any Cause Through Day 28- Modified Intent-To-Treat (mITT) Population
Description: Percentage of participants with COVID-19 related hospitalization or death from any cause during the first 28 days of the study was estimated using the Kaplan-Meier (KM) method. Using KM method, survival probability for each time interval was calculated as the number of participants surviving divided by the number of participants at risk. Participants who had the event, dropped out, or moved out were not counted as "at risk" i.e., participants who were lost were considered "censored" and were not counted in the denominator.
Time Frame: From Day 1 to Day 28
Population: mITT population included all participants who were randomized and took at least one dose of study intervention, who at baseline did not receive nor were expected to receive COVID-19 therapeutic monoclonal antibody (mAb) treatment and were treated <=3 days of COVID-19 onset.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | PF-07321332 300 mg + Ritonavir 100 mg | Placebo
Number analyzed (Participants) | 671 | 647
Percentage of participants | 0.752 [0.313 to 1.796] | 6.888 [5.172 to 9.146]
Statistical Analysis 1: Comparison: PF-07321332 300 mg + Ritonavir 100 mg vs Placebo; The difference of the percentage in the 2 treatment groups and its 95% confidence interval, and p-value based on Normal approximation of the data are presented; Test type: Superiority; p < 0.0001, Normal approximation; Percentage difference = -6.137, 95% CI 2-sided [-8.208 to -4.066], Standard Error of Mean 1.057

2. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a participant, temporarily associated with the use of study intervention, whether or not considered related to the study intervention. Serious adverse event (SAE) was any untoward medical occurrence that, at any dose: resulted in death; required inpatient hospitalization or prolongation of existing hospitalization; was life-threatening; resulted in persistent or significant disability/ incapacity; congenital anomaly/birth defect; a suspected transmission via a Pfizer product of an infectious agent, pathogenic or non-pathogenic and other important medical events. AEs included both SAEs and all non-SAEs. An AE was considered as TEAE if the event started on or after start date of study intervention.
Time Frame: From start of study intervention (Day 1) up to end of safety follow-up (Day 34)
Population: Safety analysis set (SAS) included all participants who received at least one dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-07321332 300 mg + Ritonavir 100 mg | Placebo
Number analyzed (Participants) | 1038 | 1053
Participants | 228 | 256

3. Secondary Outcome: Number of Participants With AEs Leading to Discontinuation and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant, temporarily associated with the use of study treatment, whether or not considered related to the study treatment. An SAE was any untoward medical occurrence that, at any dose: resulted in death; required inpatient hospitalization or prolongation of existing hospitalization; was life-threatening; resulted in persistent or significant disability/ incapacity; congenital anomaly/birth defect; a suspected transmission via a Pfizer product of an infectious agent, pathogenic or non-pathogenic and other important medical events.
Time Frame: From start of study intervention (Day 1) up to end of safety follow-up (Day 34)
Population: SAS population included all participants who were randomized and took at least one dose of investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-07321332 300 mg + Ritonavir 100 mg | Placebo
Number analyzed (Participants) | 1038 | 1053
Participants
  AEs leading to study discontinuation | 0 | 13
  SAEs | 18 | 71

4. Secondary Outcome: Percentage of Participants With Covid-19 Related Hospitalization or Death From Any Cause Through Day 28- Modified Intent-To-Treat 1 (mITT1) Population
Description: Percentage of participants with COVID-19 related hospitalization or death from any cause during the first 28 days of the study was estimated using the Kaplan-Meier method.
Time Frame: From Day 1 to Day 28
Population: mITT1 population included all participants who were randomized and took at least one dose of study intervention and who at baseline did not receive nor were expected to receive COVID-19 therapeutic mAb treatment.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | PF-07321332 300 mg + Ritonavir 100 mg | Placebo
Number analyzed (Participants) | 977 | 989
Percentage of participants | 0.933 [0.487 to 1.786] | 6.571 [5.180 to 8.318]
Statistical Analysis 1: Comparison: PF-07321332 300 mg + Ritonavir 100 mg vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, Normal approximation; Percentage difference = -5.638, 95% CI 2-sided [-7.308 to -3.967], Standard Error of Mean 0.852

5. Secondary Outcome: Time to Sustained Alleviation of All Targeted COVID-19 Signs and Symptoms Through Day 28- mITT Population
Description: Sustained alleviation of all targeted COVID-19 signs/symptoms was defined as the event occurring on the first 4 consecutive days when all symptoms scored as moderate or severe at the time of enrollment were scored as mild or absent and those scored mild or absent at the time of enrollment were scored as absent. The first day of the 4 consecutive-day period was considered date of first event. Time to sustained alleviation (event) was calculated as first event date minus first dose date plus 1, for participants with event. For participants who completed Day 28 or discontinued the study before Day 28 without sustained alleviation (censored), time was calculated as censoring date (last date on which symptom alleviation was assessed) minus first dose date plus 1 or Day 25 whichever occurred first.
Time Frame: From Day 1 (baseline) to Day 28
Population: mITT population included all participants who were randomized and took at least one dose of study intervention, who at baseline did not receive nor were expected to receive COVID-19 therapeutic mAb treatment and were treated <=3 days of COVID-19 onset. Here "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | PF-07321332 300 mg + Ritonavir 100 mg | Placebo
Number analyzed (Participants) | 666 | 645
Days | 12.00 [12.00 to 13.00] | 15.00 [13.00 to 16.00]
Statistical Analysis 1: Comparison: PF-07321332 300 mg + Ritonavir 100 mg vs Placebo; Analysis of treatment effect on time to sustained alleviation is based on Cox proportional hazard (PH) model with treatment and geographic region effects as independent variables, and baseline SARS-CoV-2 serology status and baseline viral load (<4 logarithm to base 10 [log10] copies/milliliter [mL], >=4 log10 copies/mL) as covariates; Test type: Superiority; p = 0.0003, Cox Proportional Hazard Model; Hazard Ratio (HR) = 1.294, 95% CI 2-sided [1.136 to 1.476]

6. Secondary Outcome: Time to Sustained Alleviation of All Targeted COVID-19 Signs and Symptoms Through Day 28- mITT1 Population
Description: as for outcome 5
Time Frame: From Day 1 (baseline) to Day 28
Population: mITT1 population included all participants who were randomized and took at least one dose of study intervention and who at baseline did not receive nor were expected to receive COVID-19 therapeutic mAb treatment. Here "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | PF-07321332 300 mg + Ritonavir 100 mg | Placebo
Number analyzed (Participants) | 970 | 986
Days | 13.00 [12.00 to 13.00] | 15.00 [14.00 to 16.00]
Statistical Analysis 1: Comparison: PF-07321332 300 mg + Ritonavir 100 mg vs Placebo; Analysis of treatment effect on time to sustained alleviation is based on Cox PH model with treatment and geographic region effects as independent variables, and symptom onset duration (<=3, >3), baseline SARS-CoV-2 serology status and baseline viral load (<4 log10 copies/mL, >=4 log10 copies/mL) as covariates; Test type: Superiority; p < 0.0001, Cox Proportional Hazard Model; Hazard Ratio (HR) = 1.266, 95% CI 2-sided [1.134 to 1.412]

7. Secondary Outcome: Time to Sustained Alleviation of All Targeted COVID-19 Signs and Symptoms Through Day 28- Modified Intent-to-Treat 2 (mITT2) Population
Description: as for outcome 5
Time Frame: From Day 1 (baseline) to Day 28
Population: mITT2 population included all participants who were randomized and took at least one dose of study intervention. Here "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | PF-07321332 300 mg + Ritonavir 100 mg | Placebo
Number analyzed (Participants) | 1031 | 1050
Days | 13.00 [12.00 to 13.00] | 16.00 [15.00 to 17.00]
Statistical Analysis 1: Comparison: PF-07321332 300 mg + Ritonavir 100 mg vs Placebo; Analysis of treatment effect on time to sustained alleviation is based on Cox PH model with treatment and geographic region effects as independent variables, and symptom onset duration (<=3, >3), COVID-19 mAb treatment (Yes/No), baseline SARS-CoV-2 serology status and baseline viral load (<4 log10 copies/mL, >=4 log10 copies/mL) as covariates; Test type: Superiority; p < 0.0001, Cox Proportional Hazard Model; Hazard Ratio (HR) = 1.258, 95% CI 2-sided [1.131 to 1.400]

8. Secondary Outcome: Percentage of Participants With Severe Covid-19 Signs and Symptoms Through Day 28- mITT Population
Description: Participants were required to record the severity of their Covid-19 symptoms over the past 24 hours daily on a 4-point scale ranging from 0 to 3, higher scores indicated more severity. The scale was reported as 0= no symptoms, 1=mild, 2=moderate and 3=severe. A participant with severe score for any targeted symptoms post-baseline was counted as severe. Percentage of participants with severe Covid-19 signs and symptoms were reported.
Time Frame: From Day 1 to Day 28
Population: as for outcome 5
Measure: Number; unit: Percentage of participants
Arm/Group | PF-07321332 300 mg + Ritonavir 100 mg | Placebo
Number analyzed (Participants) | 666 | 645
Percentage of participants | 18.168 | 20.775
Statistical Analysis 1: Comparison: PF-07321332 300 mg + Ritonavir 100 mg vs Placebo; Odds ratio, 95% CI and p-value were computed from a logistic regression model including main effects of treatment, geographic region, baseline SARS-CoV-2 serology status and baseline viral load (< 4 log10 copies/mL, >= 4 log10 copies/mL); Test type: Superiority; p = 0.3473, Regression, Logistic; Odds Ratio (OR) = 0.871, 95% CI 2-sided [0.652 to 1.162]

9. Secondary Outcome: Percentage of Participants With Severe Covid-19 Signs and Symptoms Through Day 28- mITT1 Population
Description: as for outcome 8
Time Frame: From Day 1 to Day 28
Population: as for outcome 6
Measure: Number; unit: Percentage of participants
Arm/Group | PF-07321332 300 mg + Ritonavir 100 mg | Placebo
Number analyzed (Participants) | 970 | 986
Percentage of participants | 19.691 | 21.298
Statistical Analysis 1: Comparison: PF-07321332 300 mg + Ritonavir 100 mg vs Placebo; Odds ratio, 95% CI and p-value were computed from a logistic regression model including main effects of treatment, geographic region, symptom onset duration (<=3, >3), baseline SARS-CoV-2 serology status and baseline viral load (< 4 log10 copies/mL, >= 4 log10 copies/mL); Test type: Superiority; p = 0.5762, Regression, Logistic; Odds Ratio (OR) = 0.936, 95% CI 2-sided [0.740 to 1.182]

10. Secondary Outcome: Percentage of Participants With Severe Covid-19 Signs and Symptoms Through Day 28- mITT2 Population
Description: as for outcome 8
Time Frame: From Day 1 to Day 28
Population: as for outcome 7
Measure: Number; unit: Percentage of participants
Arm/Group | PF-07321332 300 mg + Ritonavir 100 mg | Placebo
Number analyzed (Participants) | 1031 | 1050
Percentage of participants | 20.660 | 21.810
Statistical Analysis 1: Comparison: PF-07321332 300 mg + Ritonavir 100 mg vs Placebo; Odds ratio, 95% CI and p-value were computed from a logistic regression model including main effects of treatment, geographic region, symptom onset duration (<=3, >3), COVID-19 mAb treatment (Yes/No),baseline SARS-CoV-2 serology status and baseline viral load (< 4 log10 copies/mL, >= 4 log10 copies/mL); Test type: Superiority; p = 0.7807, Regression, Logistic; Odds Ratio (OR) = 0.969, 95% CI 2-sided [0.773 to 1.213]

11. Secondary Outcome: Time to Sustained Resolution of All Targeted COVID-19 Signs and Symptoms Through Day 28- mITT Population
Description: Sustained resolution was defined as when all targeted symptoms were scored as absent for 4 consecutive days. Time to sustained resolution (event) was calculated as first event date minus first dose date plus 1, for participants with event. For participants who completed Day 28 or discontinued the study before Day 28 without sustained resolution (censored), time was calculated as censoring date (last date on which symptom resolution was assessed) minus first dose date plus 1 or Day 25 whichever occurred first.
Time Frame: From Day 1 (baseline) to Day 28
Population: as for outcome 5
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | PF-07321332 300 mg + Ritonavir 100 mg | Placebo
Number analyzed (Participants) | 671 | 647
Days | 16.00 [15.00 to 17.00] | 18.00 [17.00 to 20.00]
Statistical Analysis 1: Comparison: PF-07321332 300 mg + Ritonavir 100 mg vs Placebo; Analysis of treatment effect on time to sustained resolution is based on Cox PH model with treatment and geographic region effects as independent variables, and baseline SARS-CoV-2 serology status and baseline viral load (<4 log10 copies/mL, >=4 log10 copies/mL) as covariates; Test type: Superiority; p = 0.0053, Cox Proportional Hazard Model; Hazard Ratio (HR) = 1.219, 95% CI 2-sided [1.061 to 1.401]

12. Secondary Outcome: Time to Sustained Resolution of All Targeted COVID-19 Signs and Symptoms Through Day 28- mITT1 Population
Description: as for outcome 11
Time Frame: From Day 1 (baseline) to Day 28
Population: as for outcome 6
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | PF-07321332 300 mg + Ritonavir 100 mg | Placebo
Number analyzed (Participants) | 977 | 989
Days | 16.00 [15.00 to 18.00] | 19.00 [18.00 to 20.00]
Statistical Analysis 1: Comparison: PF-07321332 300 mg + Ritonavir 100 mg vs Placebo; Analysis of treatment effect on time to sustained resolution is based on Cox PH model with treatment and geographic region effects as independent variables, and symptom onset duration (<=3, >3), baseline SARS-CoV-2 serology status and baseline viral load (<4 log10 copies/mL, >=4 log10 copies/mL) as covariates; Test type: Superiority; p = 0.0022, Cox Proportional Hazard Model; Hazard Ratio (HR) = 1.200, 95% CI 2-sided [1.068 to 1.348]

13. Secondary Outcome: Time to Sustained Resolution of All Targeted COVID-19 Signs and Symptoms Through Day 28- mITT2 Population
Description: as for outcome 11
Time Frame: From Day 1 (baseline) to Day 28
Population: as for outcome 7
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | PF-07321332 300 mg + Ritonavir 100 mg | Placebo
Number analyzed (Participants) | 1038 | 1053
Days | 17.00 [15.00 to 18.00] | 19.00 [18.00 to 20.00]
Statistical Analysis 1: Comparison: PF-07321332 300 mg + Ritonavir 100 mg vs Placebo; Analysis of treatment effect on time to sustained resolution is based on Cox PH model with treatment and geographic region effects as independent variables, and symptom onset duration (<=3, >3), COVID-19 mAb treatment (Yes/No), baseline SARS-CoV-2 serology status and baseline viral load (<4 log10 copies/mL, >=4 log10 copies/mL) as covariates; Test type: Superiority; p = 0.0021, Cox Proportional Hazard Model; Hazard Ratio (HR) = 1.194, 95% CI 2-sided [1.066 to 1.337]

14. Secondary Outcome: Time to Sustained Alleviation of Each Targeted COVID-19 Signs and Symptoms- mITT Population
Description: Sustained alleviation of each targeted COVID-19 signs/symptoms was defined as the event occurring on the first 4 consecutive days when each symptom scored as moderate or severe at the time of enrollment were scored as mild or absent and those scored mild or absent at the time of enrollment were scored as absent. The first day of the 4 consecutive-day period was considered date of first event. Time to sustained alleviation (event) was calculated as first event date minus first dose date plus 1, for participants with event. For participants who completed Day 28 or discontinued the study before Day 28 without sustained alleviation (censored), time was calculated as censoring date (last date on which symptom alleviation was assessed) minus first dose date plus 1 or Day 25 whichever occurred first.
Time Frame: From Day 1 (baseline) to Day 28
Population: mITT population included all participants who were randomized and took at least one dose of study intervention, who at baseline did not receive nor were expected to receive COVID-19 therapeutic mAb treatment and were treated <=3 days of COVID-19 onset. Here "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure. Here, "Number Analyzed" signifies participants evaluable for each specified category.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | PF-07321332 300 mg + Ritonavir 100 mg | Placebo
Number analyzed (Participants) | 671 | 647
Days
  Muscle or body aches: number analyzed (Participants) | 528 | 506
  Muscle or body aches | 6.000 [5.000 to 7.000] | 7.000 [6.000 to 8.000]
  Shortness of breath or difficulty breathing: number analyzed (Participants) | 277 | 290
  Shortness of breath or difficulty breathing | 6.000 [5.000 to 7.000] | 8.000 [6.000 to 9.000]
  Chills or shivering: number analyzed (Participants) | 412 | 376
  Chills or shivering | 3.000 [3.000 to 4.000] | 5.000 [4.000 to 5.000]
  Cough: number analyzed (Participants) | 539 | 525
  Cough | 8.000 [8.000 to 9.000] | 10.000 [9.000 to 11.000]
  Diarrhea: number analyzed (Participants) | 165 | 143
  Diarrhea | 4.000 [3.000 to 6.000] | 4.000 [3.000 to 6.000]
  Feeling hot or feverish: number analyzed (Participants) | 420 | 398
  Feeling hot or feverish | 3.000 [3.000 to 4.000] | 5.000 [4.000 to 5.000]
  Headache: number analyzed (Participants) | 494 | 453
  Headache | 5.000 [4.000 to 5.000] | 7.000 [6.000 to 8.000]
  Nausea: number analyzed (Participants) | 221 | 220
  Nausea | 4.000 [3.000 to 5.000] | 5.000 [4.000 to 7.000]
  Stuffy or runny nose: number analyzed (Participants) | 466 | 440
  Stuffy or runny nose | 6.000 [5.000 to 7.000] | 7.000 [7.000 to 8.000]
  Sore throat: number analyzed (Participants) | 373 | 347
  Sore throat | 5.000 [4.000 to 5.000] | 6.000 [5.000 to 7.000]
  Vomit: number analyzed (Participants) | 69 | 70
  Vomit | 3.000 [2.000 to 4.000] | 3.000 [2.000 to 5.000]

15. Secondary Outcome: Time to Sustained Alleviation of Each Targeted COVID-19 Signs and Symptoms- mITT1 Population
Description: as for outcome 14
Time Frame: From Day 1 (baseline) to Day 28
Population: mITT1 population included all participants who were randomized and took at least one dose of study intervention and who at baseline did not receive nor were expected to receive COVID-19 therapeutic mAb treatment. Here "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure. Here, "Number Analyzed" signifies participants evaluable for each specified category.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | PF-07321332 300 mg + Ritonavir 100 mg | Placebo
Number analyzed (Participants) | 977 | 989
Days
  Muscle or body aches: number analyzed (Participants) | 772 | 778
  Muscle or body aches | 6.000 [5.000 to 7.000] | 7.000 [7.000 to 8.000]
  Shortness of breath or difficulty breathing: number analyzed (Participants) | 423 | 451
  Shortness of breath or difficulty breathing | 6.000 [5.000 to 7.000] | 8.000 [7.000 to 10.000]
  Chills or shivering: number analyzed (Participants) | 584 | 578
  Chills or shivering | 3.000 [3.000 to 4.000] | 5.000 [4.000 to 5.000]
  Cough: number analyzed (Participants) | 791 | 816
  Cough | 9.000 [8.000 to 9.000] | 10.000 [9.000 to 11.000]
  Diarrhea: number analyzed (Participants) | 262 | 246
  Diarrhea | 5.000 [4.000 to 6.000] | 4.000 [3.000 to 5.000]
  Feeling hot or feverish: number analyzed (Participants) | 603 | 613
  Feeling hot or feverish | 3.000 [3.000 to 4.000] | 5.000 [4.000 to 6.000]
  Headache: number analyzed (Participants) | 709 | 709
  Headache | 5.000 [5.000 to 6.000] | 7.000 [7.000 to 8.000]
  Nausea: number analyzed (Participants) | 348 | 363
  Nausea | 5.000 [4.000 to 6.000] | 6.000 [5.000 to 7.000]
  Stuffy or runny nose: number analyzed (Participants) | 690 | 684
  Stuffy or runny nose | 6.000 [5.000 to 7.000] | 7.000 [7.000 to 8.000]
  Sore throat: number analyzed (Participants) | 548 | 560
  Sore throat | 5.000 [4.000 to 5.000] | 6.000 [5.000 to 7.000]
  Vomit: number analyzed (Participants) | 116 | 115
  Vomit | 3.000 [2.000 to 4.000] | 3.000 [2.000 to 5.000]

16. Secondary Outcome: Time to Sustained Alleviation of Each Targeted COVID-19 Signs and Symptoms- mITT2 Population
Description: as for outcome 14
Time Frame: From Day 1 (baseline) to Day 28
Population: mITT2 population included all participants who were randomized and took at least one dose of study intervention. Here "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure. Here, "Number Analyzed" signifies participants evaluable for each specified category.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | PF-07321332 300 mg + Ritonavir 100 mg | Placebo
Number analyzed (Participants) | 1038 | 1053
Days
  Muscle or body aches: number analyzed (Participants) | 821 | 830
  Muscle or body aches | 6.000 [6.000 to 7.000] | 8.000 [7.000 to 9.000]
  Shortness of breath or difficulty breathing: number analyzed (Participants) | 459 | 487
  Shortness of breath or difficulty breathing | 6.000 [5.000 to 7.000] | 9.000 [8.000 to 10.000]
  Chills or shivering: number analyzed (Participants) | 627 | 620
  Chills or shivering | 3.000 [3.000 to 4.000] | 5.000 [4.000 to 5.000]
  Cough: number analyzed (Participants) | 843 | 874
  Cough | 9.000 [8.000 to 9.000] | 10.000 [9.000 to 11.000]
  Diarrhea: number analyzed (Participants) | 287 | 276
  Diarrhea | 5.000 [4.000 to 6.000] | 4.000 [3.000 to 5.000]
  Feeling hot or feverish: number analyzed (Participants) | 649 | 656
  Feeling hot or feverish | 3.000 [3.000 to 4.000] | 5.000 [4.000 to 5.000]
  Headache: number analyzed (Participants) | 759 | 760
  Headache | 5.000 [5.000 to 6.000] | 7.000 [7.000 to 8.000]
  Nausea: number analyzed (Participants) | 374 | 390
  Nausea | 5.000 [4.000 to 6.000] | 6.000 [5.000 to 7.000]
  Stuffy or runny nose: number analyzed (Participants) | 739 | 738
  Stuffy or runny nose | 6.000 [5.000 to 7.000] | 7.000 [7.000 to 8.000]
  Sore throat: number analyzed (Participants) | 582 | 607
  Sore throat | 5.000 [4.000 to 5.000] | 6.000 [5.000 to 7.000]
  Vomit: number analyzed (Participants) | 132 | 135
  Vomit | 3.000 [3.000 to 4.000] | 3.000 [2.000 to 5.000]

17. Secondary Outcome: Time to Sustained Resolution of Each Targeted COVID-19 Signs and Symptoms- mITT Population
Description: Sustained resolution was defined as when each targeted symptom was scored as absent for 4 consecutive days. Time to sustained resolution (event) was calculated as first event date minus first dose date plus 1, for participants with event. For participants who completed Day 28 or discontinued the study before Day 28 without sustained resolution (censored), time was calculated as censoring date (last date on which symptom resolution was assessed) minus first dose date plus 1 or Day 25 whichever occurred first.
Time Frame: From Day 1 (baseline) to Day 28
Population: as for outcome 14
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | PF-07321332 300 mg + Ritonavir 100 mg | Placebo
Number analyzed (Participants) | 671 | 647
Days
  Muscle or body aches: number analyzed (Participants) | 528 | 506
  Muscle or body aches | 9.000 [8.000 to 11.000] | 12.000 [11.000 to 13.000]
  Shortness of breath or difficulty breathing: number analyzed (Participants) | 227 | 290
  Shortness of breath or difficulty breathing | 8.000 [7.000 to 9.000] | 11.000 [10.000 to 14.000]
  Chills or shivering: number analyzed (Participants) | 412 | 376
  Chills or shivering | 5.000 [4.000 to 5.000] | 7.000 [6.000 to 8.000]
  Cough: number analyzed (Participants) | 539 | 525
  Cough | 13.000 [12.000 to 13.000] | 15.000 [14.000 to 16.000]
  Diarrhea: number analyzed (Participants) | 165 | 143
  Diarrhea | 6.000 [5.000 to 8.000] | 6.000 [4.000 to 9.000]
  Feeling hot or feverish: number analyzed (Participants) | 420 | 398
  Feeling hot or feverish | 5.000 [4.000 to 5.000] | 7.000 [6.000 to 8.000]
  Headache: number analyzed (Participants) | 494 | 453
  Headache | 8.000 [8.000 to 9.000] | 11.000 [9.000 to 12.000]
  Nausea: number analyzed (Participants) | 221 | 220
  Nausea | 5.000 [4.000 to 7.000] | 7.000 [6.000 to 10.000]
  Stuffy or runny nose: number analyzed (Participants) | 466 | 440
  Stuffy or runny nose | 9.000 [9.000 to 10.000] | 10.000 [9.000 to 11.000]
  Sore throat: number analyzed (Participants) | 373 | 347
  Sore throat | 7.000 [6.000 to 7.000] | 9.000 [8.000 to 10.000]
  Vomit: number analyzed (Participants) | 69 | 70
  Vomit | 3.000 [2.000 to 5.000] | 3.000 [2.000 to 5.000]

18. Secondary Outcome: Time to Sustained Resolution of Each Targeted COVID-19 Signs and Symptoms- mITT1 Population
Description: as for outcome 17
Time Frame: From Day 1 (baseline) to Day 28
Population: as for outcome 15
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | PF-07321332 300 mg + Ritonavir 100 mg | Placebo
Number analyzed (Participants) | 977 | 989
Days
  Muscle or body aches: number analyzed (Participants) | 772 | 778
  Muscle or body aches | 9.000 [8.000 to 10.000] | 12.000 [11.000 to 13.000]
  Shortness of breath or difficulty breathing: number analyzed (Participants) | 423 | 451
  Shortness of breath or difficulty breathing | 9.000 [8.000 to 10.000] | 12.000 [11.000 to 15.000]
  Chills or shivering: number analyzed (Participants) | 548 | 578
  Chills or shivering | 5.000 [4.000 to 5.000] | 7.000 [6.000 to 8.000]
  Cough: number analyzed (Participants) | 791 | 816
  Cough | 13.000 [12.000 to 14.000] | 15.000 [14.000 to 17.000]
  Diarrhea: number analyzed (Participants) | 262 | 246
  Diarrhea | 6.000 [6.000 to 8.000] | 6.000 [5.000 to 8.000]
  Feeling hot or feverish: number analyzed (Participants) | 603 | 613
  Feeling hot or feverish | 5.000 [NA to NA] — Due to variability of data, the number of participants with events available was not sufficient for the calculation of the limits using KM. | 7.000 [6.000 to 8.000]
  Headache: number analyzed (Participants) | 709 | 709
  Headache | 9.000 [8.000 to 10.000] | 11.000 [10.000 to 13.000]
  Nausea: number analyzed (Participants) | 348 | 363
  Nausea | 7.000 [6.000 to 8.000] | 7.000 [6.000 to 9.000]
  Stuffy or runny nose: number analyzed (Participants) | 690 | 684
  Stuffy or runny nose | 9.000 [9.000 to 10.000] | 10.000 [9.000 to 11.000]
  Sore throat: number analyzed (Participants) | 548 | 560
  Sore throat | 7.000 [6.000 to 8.000] | 9.000 [8.000 to 10.000]
  Vomit: number analyzed (Participants) | 116 | 115
  Vomit | 3.000 [3.000 to 5.000] | 3.000 [2.000 to 5.000]

19. Secondary Outcome: Time to Sustained Resolution of Each Targeted COVID-19 Signs and Symptoms- mITT2 Population
Description: as for outcome 17
Time Frame: From Day 1 (baseline) to Day 28
Population: as for outcome 16
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | PF-07321332 300 mg + Ritonavir 100 mg | Placebo
Number analyzed (Participants) | 1038 | 1053
Days
  Muscle or body aches: number analyzed (Participants) | 821 | 830
  Muscle or body aches | 9.000 [8.000 to 10.000] | 12.000 [11.000 to 13.000]
  Shortness of breath or difficulty breathing: number analyzed (Participants) | 459 | 487
  Shortness of breath or difficulty breathing | 9.000 [8.000 to 10.000] | 13.000 [11.000 to 15.000]
  Chills or shivering: number analyzed (Participants) | 627 | 620
  Chills or shivering | 5.000 [4.000 to 5.000] | 7.000 [6.000 to 8.000]
  Cough: number analyzed (Participants) | 843 | 872
  Cough | 13.000 [12.000 to 14.000] | 15.000 [14.000 to 17.000]
  Diarrhea: number analyzed (Participants) | 287 | 276
  Diarrhea | 6.000 [6.000 to 8.000] | 6.000 [5.000 to 8.000]
  Feeling hot or feverish: number analyzed (Participants) | 649 | 656
  Feeling hot or feverish | 5.000 [5.000 to 6.000] | 7.000 [6.000 to 8.000]
  Headache: number analyzed (Participants) | 759 | 760
  Headache | 9.000 [9.000 to 10.000] | 11.000 [10.000 to 13.000]
  Nausea: number analyzed (Participants) | 374 | 390
  Nausea | 7.000 [6.000 to 8.000] | 7.000 [6.000 to 9.000]
  Stuffy or runny nose: number analyzed (Participants) | 739 | 738
  Stuffy or runny nose | 9.000 [9.000 to 10.000] | 11.000 [10.000 to 12.000]
  Sore throat: number analyzed (Participants) | 584 | 607
  Sore throat | 7.000 [6.000 to 8.000] | 9.000 [8.000 to 10.000]
  Vomit: number analyzed (Participants) | 132 | 135
  Vomit | 3.000 [3.000 to 5.000] | 4.000 [3.000 to 5.000]

20. Secondary Outcome: Number of Participants With Progression to a Worsening Status in 1 or More Self-reported COVID-19 Associated Symptoms Through Day 28-mITT Population
Description: Participants were required to record the severity of their Covid-19 symptoms over the past 24 hours daily on a 4-point scale where 0 = no symptoms; 1= mild; 2= moderate; and 3= severe. Vomiting and diarrhea were each rated on a 4-point frequency scale where 0= no occurrence, 1= mild for 1 to 2 times, 2= moderate for 3 to 4 times, and 3= severe for 5 or greater. Progression to a worsening status for any targeted symptom was based up on increasing severity (i.e. the first time any targeted symptoms worsened after treatment relative to baseline).
Time Frame: From Day 1 (baseline) to Day 28
Population: mITT population included all participants who were randomized and took at least one dose of study intervention, who at baseline did not receive nor were expected to receive COVID-19 therapeutic mAb treatment and were treated <=3 days of COVID-19 onset. Here 'Overall Number of Participants Analyzed' signifies participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-07321332 300 mg + Ritonavir 100 mg | Placebo
Number analyzed (Participants) | 666 | 645
Participants | 507 | 483
Statistical Analysis 1: Comparison: PF-07321332 300 mg + Ritonavir 100 mg vs Placebo; [analysis description as in outcome 8, analysis 1]; Test type: Superiority; p = 0.5293, Regression, Logistic; Odds Ratio (OR) = 1.088, 95% CI 2-sided [0.836 to 1.416]

21. Secondary Outcome: Number of Participants With Progression to a Worsening Status in 1 or More Self-reported COVID-19 Associated Symptoms Through Day 28-mITT1 Population
Description: as for outcome 20
Time Frame: From Day 1 (baseline) to Day 28
Population: mITT1 population included all participants who were randomized and took at least one dose of study intervention and who at baseline did not receive nor were expected to receive COVID-19 therapeutic mAb treatment. Here 'Overall Number of Participants Analyzed' signifies participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-07321332 300 mg + Ritonavir 100 mg | Placebo
Number analyzed (Participants) | 970 | 986
Participants | 735 | 737
Statistical Analysis 1: Comparison: PF-07321332 300 mg + Ritonavir 100 mg vs Placebo; [analysis description as in outcome 9, analysis 1]; Test type: Superiority; p = 0.6379, Regression, Logistic; Odds Ratio (OR) = 1.053, 95% CI 2-sided [0.850 to 1.303]

22. Secondary Outcome: Number of Participants With Progression to a Worsening Status in 1 or More Self-reported COVID-19 Associated Symptoms Through Day 28-mITT2 Population
Description: as for outcome 20
Time Frame: From Day 1 (baseline) to Day 28
Population: mITT2 population included all participants who were randomized and took at least one dose of study intervention. Here 'Overall Number of Participants Analyzed' signifies participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-07321332 300 mg + Ritonavir 100 mg | Placebo
Number analyzed (Participants) | 1031 | 1050
Participants | 787 | 790
Statistical Analysis 1: Comparison: PF-07321332 300 mg + Ritonavir 100 mg vs Placebo; Odds ratio, 95% CI and p-value were computed from a logistic regression model including main effects of treatment, geographic region, symptom onset duration (<=3, >3), COVID-19 mAb treatment (Yes/No), baseline SARS-CoV-2 serology status and baseline viral load (< 4 log10 copies/mL, >= 4 log10 copies/mL); Test type: Superiority; p = 0.6760, Regression, Logistic; Odds Ratio (OR) = 1.046, 95% CI 2-sided [0.848 to 1.290]

23. Secondary Outcome: Percentage of Participants With a Resting Peripheral Oxygen Saturation >=95% at Days 1 and 5- mITT Population
Description: In this outcome measure, the percentage of participants with a resting peripheral oxygen saturation >=95% were reported.
Time Frame: Day 1, 5
Population: mITT population included all participants who were randomized and took at least one dose of study intervention, who at baseline did not receive nor were expected to receive COVID-19 therapeutic mAb treatment and were treated <=3 days of COVID-19 onset. Here, "Number Analyzed" signifies participants evaluable for each specified timepoint.
Measure: Number; unit: Percentage of participants
Arm/Group | PF-07321332 300 mg + Ritonavir 100 mg | Placebo
Number analyzed (Participants) | 671 | 647
Percentage of participants
  Day 1 | 93.443 | 91.963
  Day 5: number analyzed (Participants) | 627 | 595
  Day 5 | 92.823 | 89.076
Statistical Analysis 1: Comparison: PF-07321332 300 mg + Ritonavir 100 mg vs Placebo; Test type: Superiority; p = 0.1997, Breslow-Day test; Odds Ratio (OR) = 19.400, 95% CI [7.788 to 48.328] — Odds ratio for Day 5 vs Day 1: PF-07321332 300 mg + Ritonavir 100 mg
Statistical Analysis 2: Comparison: PF-07321332 300 mg + Ritonavir 100 mg vs Placebo; Test type: Other; Breslow-Day test; Odds Ratio (OR) = 8.948, 95% CI 2-sided [4.159 to 19.253] — Odds ratio for Day 5 vs Day 1: Placebo

24. Secondary Outcome: Percentage of Participants With a Resting Peripheral Oxygen Saturation >=95% at Days 1 and 5- mITT1 Population
Description: In this outcome measure, the percentage of participants with a resting peripheral oxygen saturation >=95% were reported.
Time Frame: Day 1, 5
Population: mITT1 population included all participants who were randomized and took at least one dose of study intervention and who at baseline did not receive nor were expected to receive COVID-19 therapeutic mAb treatment. Here, "Number Analyzed" signifies participants evaluable for each specified time point.
Measure: Number; unit: Percentage of participants
Arm/Group | PF-07321332 300 mg + Ritonavir 100 mg | Placebo
Number analyzed (Participants) | 977 | 989
Percentage of participants
  Day 1 | 93.347 | 92.214
  Day 5: number analyzed (Participants) | 912 | 912
  Day 5 | 91.577 | 87.610
Statistical Analysis 1: Comparison: PF-07321332 300 mg + Ritonavir 100 mg vs Placebo; Test type: Superiority; p = 0.2810, Breslow-Day test; Odds Ratio (OR) = 20.875, 95% CI 2-sided [10.097 to 43.156] — Odds ratio for Day 5 vs Day 1: PF-07321332 300 mg + Ritonavir 100 mg
Statistical Analysis 2: Comparison: PF-07321332 300 mg + Ritonavir 100 mg vs Placebo; Test type: Superiority; Breslow Day test; Odds Ratio (OR) = 12.452, 95% CI 2-sided [6.823 to 22.725] — Odds ratio for Day 5 vs Day 1: Placebo

25. Secondary Outcome: Percentage of Participants With a Resting Peripheral Oxygen Saturation >=95% at Days 1 and 5- mITT2 Population
Description: In this outcome measure, the percentage of participants with a resting peripheral oxygen saturation >=95% were reported.
Time Frame: Day 1, 5
Population: mITT2 population included all participants who were randomized and took at least one dose of study intervention. Here, "Number Analyzed" signifies participants evaluable for each specified time point.
Measure: Number; unit: Percentage of participants
Arm/Group | PF-07321332 300 mg + Ritonavir 100 mg | Placebo
Number analyzed (Participants) | 1038 | 1053
Percentage of participants
  Day 1 | 93.353 | 91.738
  Day 5: number analyzed (Participants) | 969 | 966
  Day 5 | 91.538 | 87.681
Statistical Analysis 1: Comparison: PF-07321332 300 mg + Ritonavir 100 mg vs Placebo; Test type: Superiority; p = 0.2226, Breslow-Day test; Odds Ratio (OR) = 21.119, 95% CI 2-sided [10.412 to 42.837] — Odds ratio for Day 5 vs Day 1: PF-07321332 300 mg + Ritonavir 100 mg
Statistical Analysis 2: Comparison: PF-07321332 300 mg + Ritonavir 100 mg vs Placebo; Test type: Superiority; p = 0.2342, Breslow-Day test; Odds Ratio (OR) = 12.036, 95% CI 2-sided [6.808 to 21.280] — Odds ratio for Day 5 vs Day 1: Placebo

26. Secondary Outcome: Percentage of Participants Who Died Through Week 24- mITT Population
Description: In this outcome measure, percentage of participants with death due to any cause was presented.
Time Frame: From Day 1 up to Week 24
Population: mITT population included all participants who were randomized and took at least one dose of study intervention, who at baseline did not receive nor were expected to receive COVID-19 therapeutic mAb treatment and were treated <=3 days of COVID-19 onset.
Measure: Number; unit: Percentage of participants
Arm/Group | PF-07321332 300 mg + Ritonavir 100 mg | Placebo
Number analyzed (Participants) | 671 | 647
Percentage of participants | 0 | 1.7

27. Secondary Outcome: Percentage of Participants Who Died Through Week 24- mITT1 Population
Description: In this outcome measure, percentage of participants with death due to any cause was presented.
Time Frame: From Day 1 up to Week 24
Population: as for outcome 4
Measure: Number; unit: Percentage of participants
Arm/Group | PF-07321332 300 mg + Ritonavir 100 mg | Placebo
Number analyzed (Participants) | 977 | 989
Percentage of participants | 0 | 1.5

28. Secondary Outcome: Percentage of Participants Who Died Through Week 24- mITT2 Population
Description: In this outcome measure, percentage of participants with death due to any cause was presented.
Time Frame: From Day 1 up to Week 24
Population: mITT2 population included all participants who were randomized and took at least one dose of study intervention.
Measure: Number; unit: Percentage of participants
Arm/Group | PF-07321332 300 mg + Ritonavir 100 mg | Placebo
Number analyzed (Participants) | 1038 | 1053
Percentage of participants | 0 | 1.4

29. Secondary Outcome: Plasma Concentration Versus Time Summary of PF-07321332
Time Frame: 1 Hour post-dose on Day 1 and pre-dose on Day 5
Population: SAS population included all participants who were randomized and took at least one dose of study intervention. Here "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure. Here "Number Analyzed" signifies participants evaluable for the specified time point.
Measure: Mean (Standard Deviation); unit: Nanograms per milliliter
Arm/Group | PF-07321332 300 mg + Ritonavir 100 mg
Number analyzed (Participants) | 772
Nanograms per milliliter
  Day 1 (1 Hour post dose): number analyzed (Participants) | 267
  Day 1 (1 Hour post dose) | 2201 (2130.7)
  Day 5 (Pre-dose): number analyzed (Participants) | 505
  Day 5 (Pre-dose) | 3087 (2884.3)

30. Secondary Outcome: Change From Baseline in Logarithm to Base10 (Log10) Transformed Viral Load at Day 3, 5, 10 and 14- mITT Population
Description: The viral load was measured in nasal or nasopharyngeal samples using reverse transcription polymerase chain reaction (RT-PCR).
Time Frame: Baseline, Day 3, 5, 10 and 14
Population: mITT population included all participants who were randomized and took at least one dose of study intervention, who at baseline did not receive nor were expected to receive COVID-19 therapeutic mAb treatment and were treated <=3 days of COVID-19 onset. Here "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure. Here, "Number Analyzed" signifies participants evaluable for each specified time point.
Measure: Mean (Standard Deviation); unit: Log10 copies per milliliter
Arm/Group | PF-07321332 300 mg + Ritonavir 100 mg | Placebo
Number analyzed (Participants) | 671 | 647
Log10 copies per milliliter
  Day 3: number analyzed (Participants) | 509 | 498
  Day 3 | -1.829 (1.805) | -1.203 (1.697)
  Day 5: number analyzed (Participants) | 487 | 478
  Day 5 | -3.244 (1.697) | -2.923 (1.787)
  Day 10: number analyzed (Participants) | 482 | 447
  Day 10 | -4.522 (2.105) | -3.964 (2.1115)
  Day 14: number analyzed (Participants) | 486 | 472
  Day 14 | -5.108 (2.141) | -4.862 (2.121)

31. Secondary Outcome: Change From Baseline in Log10 Transformed Viral Load at Day 3, 5, 10 and 14- mITT1 Population
Description: The viral load was measured in nasal or nasopharyngeal samples using RT-PCR.
Time Frame: Baseline, Day 3, 5, 10 and 14
Population: mITT1 population included all participants who were randomized and took at least one dose of study intervention and who at baseline did not receive nor were expected to receive COVID-19 therapeutic mAb treatment. Here "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure. Here, "Number Analyzed" signifies participants evaluable for each specified time point.
Measure: Mean (Standard Deviation); unit: Log10 copies per milliliter
Arm/Group | PF-07321332 300 mg + Ritonavir 100 mg | Placebo
Number analyzed (Participants) | 977 | 989
Log10 copies per milliliter
  Day 3: number analyzed (Participants) | 718 | 733
  Day 3 | -1.790 (1.727) | -1.182 (1.689)
  Day 5: number analyzed (Participants) | 688 | 694
  Day 5 | -3.064 (1.708) | -2.213 (1.754)
  Day 10: number analyzed (Participants) | 682 | 663
  Day 10 | -4.309 (2.108) | -3.772 (2.058)
  Day 14: number analyzed (Participants) | 691 | 698
  Day 14 | -4.878 (2.144) | -4.556 (2.146)

32. Secondary Outcome: Change From Baseline in Log10 Transformed Viral Load at Day 3, 5, 10 and 14- mITT2 Population
Description: The viral load was measured in nasal or nasopharyngeal samples using RT-PCR.
Time Frame: Baseline, Day 3, 5, 10 and 14
Population: mITT2 population included all participants who were randomized and took at least one dose of study intervention. Here 'Overall Number of Participants Analyzed' signifies participants evaluable for this outcome measure. Here, "Number Analyzed" signifies participants evaluable for each specified time point.
Measure: Mean (Standard Deviation); unit: Log10 copies per milliliter
Arm/Group | PF-07321332 300 mg + Ritonavir 100 mg | Placebo
Number analyzed (Participants) | 1038 | 1053
Log10 copies per milliliter
  Day 3: number analyzed (Participants) | 766 | 781
  Day 3 | -1.828 (1.715) | -1.178 (1.663)
  Day 5: number analyzed (Participants) | 735 | 743
  Day 5 | -3.097 (1.692) | -2.239 (1.741)
  Day 10: number analyzed (Participants) | 728 | 712
  Day 10 | -4.322 (2.109) | -3.777 (2.041)
  Day 14: number analyzed (Participants) | 739 | 752
  Day 14 | -4.882 (2.142) | -4.547 (2.146)

33. Secondary Outcome: Number of COVID-19 Related Medical Visits- mITT Population
Description: Medical visits included emergency room, practitioner's office, home healthcare services, urgent care, telephone consultation, outpatient infusion center, other, COVID-19-related-hospitalization (intensive care unit [ICU] and non-ICU stays). In this outcome measure, COVID-19-related medical visits of participants were reported.
Time Frame: From Day 1 up to Day 34
Population: as for outcome 26
Measure: Number; unit: Visits
Arm/Group | PF-07321332 300 mg + Ritonavir 100 mg | Placebo
Number analyzed (Participants) | 671 | 647
Visits | 22 | 81

34. Secondary Outcome: Number of COVID-19 Related Medical Visits- mITT1 Population
Description: Medical visits included emergency room, practitioner's office, home healthcare services, urgent care, telephone consultation, outpatient infusion center, other, COVID-19-related-hospitalization (ICU and non-ICU stays). In this outcome measure, COVID-19-related medical visits of participants were reported.
Time Frame: From Day 1 up to Day 34
Population: as for outcome 4
Measure: Number; unit: Visits
Arm/Group | PF-07321332 300 mg + Ritonavir 100 mg | Placebo
Number analyzed (Participants) | 977 | 989
Visits | 40 | 128

35. Secondary Outcome: Number of COVID-19 Related Medical Visits- mITT2 Population
Description: as for outcome 34
Time Frame: From Day 1 up to Day 34
Population: mITT2 population included all participants who were randomized and took at least one dose of study intervention.
Measure: Number; unit: Visits
Arm/Group | PF-07321332 300 mg + Ritonavir 100 mg | Placebo
Number analyzed (Participants) | 1038 | 1053
Visits | 45 | 144

36. Secondary Outcome: Number of Days in Hospital and ICU for the Treatment of COVID-19- mITT Population
Time Frame: From Day 1 up to Day 34
Population: mITT population included all participants who were randomized and took at least one dose of study intervention, who at baseline did not receive nor were expected to receive COVID-19 therapeutic mAb treatment and were treated <=3 days of COVID-19 onset. The analysis was performed on all participants (i.e. hospitalized and non-hospitalized participants were included).
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | PF-07321332 300 mg + Ritonavir 100 mg | Placebo
Number analyzed (Participants) | 671 | 647
Days
  Duration of hospitalization visits | 0.088 (1.049) | 0.844 (4.535)
  Duration of ICU visits | 0.000 (0.000) | 0.179 (2.389)
  Duration of non-ICU visits | 0.088 (1.049) | 0.666 (3.710)

37. Secondary Outcome: Number of Days in Hospital and ICU for the Treatment of COVID-19- mITT1 Population
Time Frame: From Day 1 up to Day 34
Population: mITT1 population included all participants who were randomized and took at least one dose of study intervention and who at baseline did not receive nor were expected to receive COVID-19 therapeutic mAb treatment. The analysis was performed on all participants (i.e. hospitalized and non-hospitalized participants were included).
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | PF-07321332 300 mg + Ritonavir 100 mg | Placebo
Number analyzed (Participants) | 977 | 989
Days
  Duration of hospitalization visits | 0.087 (0.968) | 0.766 (4.055)
  Duration of ICU visits | 0.000 (0.000) | 0.128 (1.964)
  Duration of non-ICU visits | 0.087 (0.968) | 0.639 (3.446)

38. Secondary Outcome: Number of Days in Hospital and ICU for the Treatment of COVID-19- mITT2 Population
Time Frame: From Day 1 up to Day 34
Population: mITT2 population included all participants who were randomized and took at least one dose of study intervention. The analysis was performed on all participants (i.e. hospitalized and non-hospitalized participants were included).
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | PF-07321332 300 mg + Ritonavir 100 mg | Placebo
Number analyzed (Participants) | 1038 | 1053
Days
  Duration of hospitalization visits | 0.092 (0.988) | 0.729 (3.940)
  Duration of ICU visits | 0.000 (0.000) | 0.121 (1.904)
  Duration of non-ICU visits | 0.092 (0.988) | 0.610 (3.350)

ADVERSE EVENTS:
Time Frame: From start of study intervention at Day 1 up to end of long-term safety follow-up (Week 24)
Description: Same event may appear as both non-SAE and SAE. However, what is presented are distinct events. An event may be categorized as serious in 1 participant and as non-serious in another participant, or 1 participant may have experienced both serious and non-serious event during the study. SAS population included all participants who were randomized and took at least one dose of investigational product.
Arm/Group | PF-07321332 300 mg + Ritonavir 100 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/1038 | 15/1053
Serious Adverse Events (participants affected / at risk) | 19/1038 | 72/1053
Other Adverse Events (participants affected / at risk) | 234/1038 | 228/1053
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PF-07321332 300 mg + Ritonavir 100 mg (N=1038) | Placebo (N=1053)
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Palpitations (Cardiac disorders) | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1
Chest discomfort (General disorders) | 1 | 0
Abscess (Infections and infestations) | 1 | 0
Atypical pneumonia (Infections and infestations) | 0 | 1
COVID-19 (Infections and infestations) | 2 | 7
COVID-19 pneumonia (Infections and infestations) | 7 | 36
Pneumonia (Infections and infestations) | 1 | 11
Sepsis (Infections and infestations) | 1 | 0
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 | 1
Eye injury (Injury, poisoning and procedural complications) | 0 | 1
Hand fracture (Injury, poisoning and procedural complications) | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1
Creatinine renal clearance decreased (Investigations) | 1 | 2
Fibrin D dimer increased (Investigations) | 0 | 1
Haemoglobin decreased (Investigations) | 1 | 0
Oxygen saturation decreased (Investigations) | 1 | 0
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Brain stem stroke (Nervous system disorders) | 1 | 0
Facial paralysis (Nervous system disorders) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 5
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Hypertensive crisis (Vascular disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 5
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Abortion threatened (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PF-07321332 300 mg + Ritonavir 100 mg (N=1038) | Placebo (N=1053)
Anaemia (Blood and lymphatic system disorders) | 1 | 2
Leukocytosis (Blood and lymphatic system disorders) | 2 | 0
Leukopenia (Blood and lymphatic system disorders) | 2 | 2
Lymphadenopathy mediastinal (Blood and lymphatic system disorders) | 0 | 1
Microcytic anaemia (Blood and lymphatic system disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 3
Palpitations (Cardiac disorders) | 1 | 2
Pericardial effusion (Cardiac disorders) | 0 | 1
Sinus bradycardia (Cardiac disorders) | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 1
Ventricular arrhythmia (Cardiac disorders) | 0 | 1
Hyperacusis (Ear and labyrinth disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 1
Thyroiditis chronic (Endocrine disorders) | 0 | 1
Eye pain (Eye disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 3
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 5 | 2
Aphthous ulcer (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 3
Diarrhoea (Gastrointestinal disorders) | 31 | 16
Dyspepsia (Gastrointestinal disorders) | 4 | 4
Faeces soft (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 | 1
Hiatus hernia (Gastrointestinal disorders) | 0 | 2
Hyperchlorhydria (Gastrointestinal disorders) | 0 | 1
Large intestine polyp (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 15 | 19
Toothache (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 12 | 9
Asthenia (General disorders) | 3 | 3
Catheter site pain (General disorders) | 1 | 0
Chest discomfort (General disorders) | 1 | 0
Chest pain (General disorders) | 2 | 1
Chills (General disorders) | 5 | 0
Fatigue (General disorders) | 2 | 5
Non-cardiac chest pain (General disorders) | 1 | 0
Oedema due to cardiac disease (General disorders) | 1 | 0
Pain (General disorders) | 0 | 3
Peripheral swelling (General disorders) | 0 | 1
Pyrexia (General disorders) | 8 | 7
Cholestasis (Hepatobiliary disorders) | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 2 | 1
Hepatic steatosis (Hepatobiliary disorders) | 0 | 1
Hepatitis toxic (Hepatobiliary disorders) | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0
Liver injury (Hepatobiliary disorders) | 0 | 1
Steatohepatitis (Hepatobiliary disorders) | 1 | 0
Mycotic allergy (Immune system disorders) | 1 | 0
Seasonal allergy (Immune system disorders) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 1
Bronchopulmonary aspergillosis (Infections and infestations) | 0 | 1
COVID-19 (Infections and infestations) | 7 | 7
COVID-19 pneumonia (Infections and infestations) | 1 | 6
Gastroenteritis viral (Infections and infestations) | 0 | 1
Hepatitis viral (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 0 | 1
Mumps (Infections and infestations) | 0 | 1
Nasopharyngitis (Infections and infestations) | 1 | 0
Oral candidiasis (Infections and infestations) | 0 | 1
Oral herpes (Infections and infestations) | 1 | 2
Oropharyngeal candidiasis (Infections and infestations) | 1 | 0
Pharyngitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 4
Pneumonia viral (Infections and infestations) | 0 | 1
Pyelonephritis chronic (Infections and infestations) | 1 | 0
Respiratory tract infection bacterial (Infections and infestations) | 1 | 0
Respiratory tract infection viral (Infections and infestations) | 2 | 1
Staphylococcal bacteraemia (Infections and infestations) | 0 | 1
Tonsillitis (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 1
Viral rhinitis (Infections and infestations) | 0 | 1
Viral sepsis (Infections and infestations) | 1 | 0
Vulvovaginal candidiasis (Infections and infestations) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 2
Hand fracture (Injury, poisoning and procedural complications) | 0 | 1
Ligament rupture (Injury, poisoning and procedural complications) | 0 | 1
Meniscus injury (Injury, poisoning and procedural complications) | 0 | 1
Activated partial thromboplastin time prolonged (Investigations) | 9 | 12
Alanine aminotransferase increased (Investigations) | 18 | 26
Aspartate aminotransferase increased (Investigations) | 11 | 14
Blood albumin decreased (Investigations) | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 1 | 0
Blood bicarbonate decreased (Investigations) | 1 | 1
Blood calcium decreased (Investigations) | 0 | 1
Blood calcium increased (Investigations) | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 1 | 5
Blood creatinine decreased (Investigations) | 0 | 1
Blood creatinine increased (Investigations) | 0 | 1
Blood fibrinogen decreased (Investigations) | 5 | 3
Blood glucose decreased (Investigations) | 1 | 0
Blood glucose increased (Investigations) | 1 | 7
Blood lactate dehydrogenase increased (Investigations) | 0 | 1
Blood potassium increased (Investigations) | 1 | 0
Blood pressure increased (Investigations) | 1 | 1
Blood sodium decreased (Investigations) | 0 | 2
Blood thyroid stimulating hormone decreased (Investigations) | 1 | 0
Blood thyroid stimulating hormone increased (Investigations) | 5 | 7
Blood urea increased (Investigations) | 1 | 1
Breath sounds abnormal (Investigations) | 1 | 0
C-reactive protein (Investigations) | 2 | 1
C-reactive protein increased (Investigations) | 10 | 13
Coagulation time prolonged (Investigations) | 1 | 0
Creatinine renal clearance decreased (Investigations) | 14 | 14
Creatinine renal clearance increased (Investigations) | 1 | 1
Differential white blood cell count abnormal (Investigations) | 1 | 0
Fibrin D dimer (Investigations) | 1 | 0
Fibrin D dimer increased (Investigations) | 25 | 30
Glomerular filtration rate abnormal (Investigations) | 0 | 1
Glomerular filtration rate decreased (Investigations) | 3 | 2
Glycosylated haemoglobin increased (Investigations) | 0 | 1
Haematocrit increased (Investigations) | 1 | 1
Haemoglobin decreased (Investigations) | 1 | 0
Haemoglobin increased (Investigations) | 0 | 1
Haptoglobin increased (Investigations) | 4 | 3
Hepatic enzyme abnormal (Investigations) | 0 | 1
Hepatic enzyme increased (Investigations) | 2 | 3
Hepatitis C virus test positive (Investigations) | 1 | 0
International normalised ratio abnormal (Investigations) | 1 | 0
International normalised ratio increased (Investigations) | 3 | 5
Lymphocyte count decreased (Investigations) | 0 | 3
Neutrophil count decreased (Investigations) | 0 | 2
Neutrophil count increased (Investigations) | 2 | 0
Oxygen saturation decreased (Investigations) | 0 | 1
Platelet count decreased (Investigations) | 1 | 1
Platelet count increased (Investigations) | 2 | 1
Procalcitonin increased (Investigations) | 1 | 2
Prothrombin time prolonged (Investigations) | 3 | 5
Red blood cell count increased (Investigations) | 0 | 1
Serum ferritin decreased (Investigations) | 1 | 0
Serum ferritin increased (Investigations) | 2 | 6
Thyroxine free increased (Investigations) | 0 | 1
Thyroxine increased (Investigations) | 1 | 0
Transaminases increased (Investigations) | 0 | 1
Weight increased (Investigations) | 0 | 1
White blood cell count decreased (Investigations) | 2 | 3
White blood cell count increased (Investigations) | 2 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 2 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 2 | 1
Glucose tolerance impaired (Metabolism and nutrition disorders) | 1 | 0
Gout (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 4
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 1
Hypervolaemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 3
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 1
Impaired fasting glucose (Metabolism and nutrition disorders) | 0 | 1
Lack of satiety (Metabolism and nutrition disorders) | 0 | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 3
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 2
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 7 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Amnesia (Nervous system disorders) | 0 | 1
Anosmia (Nervous system disorders) | 3 | 0
Dizziness (Nervous system disorders) | 3 | 5
Dysgeusia (Nervous system disorders) | 48 | 1
Facial paralysis (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 12 | 13
Hypersomnia (Nervous system disorders) | 0 | 1
Memory impairment (Nervous system disorders) | 1 | 0
Paraesthesia (Nervous system disorders) | 1 | 0
Parosmia (Nervous system disorders) | 1 | 0
Restless legs syndrome (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
Tension headache (Nervous system disorders) | 0 | 1
Tremor (Nervous system disorders) | 0 | 1
Vascular dementia (Nervous system disorders) | 1 | 0
Product after taste (Product Issues) | 3 | 0
Anxiety (Psychiatric disorders) | 3 | 1
Confusional state (Psychiatric disorders) | 1 | 1
Depression (Psychiatric disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 2 | 2
Stress (Psychiatric disorders) | 0 | 1
Chronic kidney disease (Renal and urinary disorders) | 1 | 2
Nephrosclerosis (Renal and urinary disorders) | 0 | 1
Renal impairment (Renal and urinary disorders) | 0 | 2
Heavy menstrual bleeding (Reproductive system and breast disorders) | 0 | 1
Intermenstrual bleeding (Reproductive system and breast disorders) | 0 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Allergic cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 6
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 | 7
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 | 0
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Acne (Skin and subcutaneous tissue disorders) | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 3
Erythema (Skin and subcutaneous tissue disorders) | 0 | 4
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 3
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 2 | 0
Skin oedema (Skin and subcutaneous tissue disorders) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 2
Disease risk factor (Social circumstances) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1
Embolism (Vascular disorders) | 0 | 2
Hyperaemia (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 8 | 4
Hypotension (Vascular disorders) | 1 | 4
Orthostatic hypotension (Vascular disorders) | 0 | 1
Thrombophlebitis (Vascular disorders) | 0 | 1
Vein collapse (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from the study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2021-11-20): https://cdn.clinicaltrials.gov/large-docs/02/NCT04960202/Prot_000.pdf
  • Statistical Analysis Plan (2022-04-28): https://cdn.clinicaltrials.gov/large-docs/02/NCT04960202/SAP_001.pdf